CLINICAL TRIAL: NCT03966014
Title: Different Duration and Dosing of Amoxicillin in Patients With Erythema Migrans. A Randomized Clinical Trial.
Brief Title: Different Amoxicillin Treatment Regimens in Erythema Migrans Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other)
Responsible Party: Principal Investigator, Daša Stupica, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Amoxy 10-15
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Erythema Migrans
MeSH Terms: conditions — Glossitis, Benign Migratory

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EM-amoxicillin 3 x 10 days (Active Comparator)
  Interventions: Drug: EM-amoxicillin 3 x 10 days
- EM-amoxicillin 3 x 14 days (Active Comparator)
  Interventions: Drug: EM-amoxicillin 3 x 14 days
- EM-amoxicillin 2 x 14 days (Active Comparator)
  Interventions: Drug: EM-amoxicillin 2 x 14 days
- Controls (Other)
  Interventions: Other: Controls

INTERVENTIONS:
Drug: EM-amoxicillin 3 x 10 days — Patients will receive amoxicillin 500 milligram tid for 10 days
  Arms: EM-amoxicillin 3 x 10 days
Drug: EM-amoxicillin 3 x 14 days — Patients will receive amoxicillin 500 milligram tid for 14 days
  Arms: EM-amoxicillin 3 x 14 days
Drug: EM-amoxicillin 2 x 14 days — Patients will receive amoxicillin 500 milligram bid for 14 days
  Arms: EM-amoxicillin 2 x 14 days
Other: Controls — No intervention.
  Arms: Controls

SUMMARY:
The purpose of this study is to compare the efficacy of different amoxicilline treatment regimens in patients with erythema migrans.

ELIGIBILITY:
Inclusion Criteria:

* erythema migrans

Exclusion Criteria:

* pregnancy
* extracutaneous manifestations of Lyme borreliosis
* immunocompromising state
* serious adverse event to beta lactam antibiotic
* receiving antibiotic with antiborrelial activity within 10 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number (frequency) of patients with objective manifestations of Lyme borreliosis or subjective Lyme borreliosis-associated/post-Lyme borreliosis symptoms | One year follow-up
  At each visit physical examination wil be performed and clinical signs indicating objective manifestations of Lyme borreliosis, such as erythema migrans, will be searched for and documented. At each visit patients will be asked an open question about any health-related symptoms that had newly developed or worsened since the onset of erythema migrans. If these symptoms will have no other known medical explanation, they will be regarded as Lyme borreliosis-associated constitutional symptoms at enrolment or post-Lyme borreliosis symptoms at follow-up.

SECONDARY OUTCOMES:
Number (frequency) of patients with nonspecific symptoms | One year follow-up
  At each visit patients will be asked to complete a written questionnaire asking whether they had had any of eight non-speciﬁc symptoms (fatigue, arthralgias, headache,myalgias, paraesthesias, memory difﬁculties, concentration difﬁculties and irritability) within the preceding week.

CONTACTS AND LOCATIONS:
Overall Officials: Daša Stupica, MD PhD, Principal Investigator — Department of Infectious Diseases, University Medical Centre Ljubljana, Slovenia
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia